CLINICAL TRIAL: NCT05661825
Title: The Efficacy and Related Factors in Phase II Cardiac Rehabilitation for the Patients With Acute Myocardial Infarction
Brief Title: Cardiac Rehabilitation for the Patients With Acute Myocardial Infarction
Status: Completed | Type: Observational
Sponsor: Taipei Medical University WanFang Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: TMU-JIRB N202207042
Record Dates: First submitted 2022-12-14; First posted 2022-12-22 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-05

CONDITIONS: Acute Myocardial Infarction
Keywords: Acute myocardial infarction; Cardiac rehabilitation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients diagnosed with acute myocardial infarction in the emergent department: The cases being admitted to the Emergent Department and than transferred to the general ward due to the diagnosis of acute myocardial infarction were included in the study (from Jan 1, 2012 to Jun 30, 2022). The age of these cases must be older than or equal to 20 years old.
  Interventions: Other: phase II cardiac rehabilitation

INTERVENTIONS:
Other: phase II cardiac rehabilitation — Phase II cardiac rehabilitation was provided in the the department of physical medicine and rehabilitation in Wan Fang Hospital. The programs are two times a week, one session for 30 minutes (30 sessions in total). The training programs are focused on aerobic training with bicycles. The training intensity is calculated with 40% to 80% oxygen consumption reserve from the result of cardiopulmonary exercise test. In case of safety, heart rate, blood pressure, EKG and rate of perceived exertion will be monitored during training.

SUMMARY:
The benefits of cardiac rehabilitation include improving exercise tolerance and quality of life. However the attending rate of the patients with acute myocardial infarction was low according to the previous studies. This is a retrospective chart review study collecting the basic characteristics of the patients diagnosed with acute myocardial infarction of Wang-Fang Hospital (from Jan 1, 2012 to June 30, 2021). The aims of the studies are to investigate the related issues of cardiac rehabilitation including (1) attending rate (2) the efficacy of exercise training (3) the factors that limit the participation of the training programs.

ELIGIBILITY:
Inclusion Criteria:

1. Cased diagnosed with acute myocardial infarction at emergent department and admitted
2. Age over 20 years old

Exclusion Criteria:

1. AAD cases after admission to ER or the general ward
2. Cases died within admission.
3. Cases refused the treatments.-

Min Age: 20 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Acute myocardial infarction
Sampling Method: Non-Probability Sample
Enrollment: 850 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2023-10-30 (Actual)

PRIMARY OUTCOMES:
Changes of maximal oxygen consumption after intervention | Baseline, 6 weeks after training, 16 weeks after training
  The subjects received cardiopulmonary exercise tests before and after training.

CONTACTS AND LOCATIONS:
Overall Officials: Shiauyee Chen, Master, Principal Investigator — Department of physical medicine and rehabilitation, Wan Fang Hospital
Locations (1):
- Wan-Fang hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No